CLINICAL TRIAL: NCT04937153
Title: Open-label, Dose-escalation Trial to Evaluate the Safety and Pharmacokinetics of GEN1046 in Japanese Subjects With Advanced Solid Malignancies
Brief Title: GEN1046 Safety and PK in Subjects With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1046-02; jRCT2031210112 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2021-05-11; First posted 2021-06-23 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: The starting dose is 15 mg administered as a flat dose. Dose escalation steps are based on safety data.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- acasunlimab monotherapy (Experimental)
  Interventions: Biological: Acasunlimab
- acasunlimab + pembrolizumab combination therapy (Experimental)
  Interventions: Biological: Acasunlimab; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Acasunlimab — Acasunlimab will be administered intravenously (IV) once every 21 days.
  Other Names: GEN1046; DuoBody®-PD-L1x4-1BB
Biological: Pembrolizumab — Pembrolizumab will be administered IV once every 21 days.
  Arms: acasunlimab + pembrolizumab combination therapy

SUMMARY:
The primary objective of the study is to evaluate the safety, tolerability, dose-limiting toxicity (DLT) and pharmacokinetics (PK) of acasunlimab (also known as GEN1046) administered as monotherapy or in combination with pembrolizumab in Japanese study participants with malignant solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant must have a histologically-confirmed non-central nervous system (CNS) solid tumor that is metastatic or unresectable and for whom there is no available standard therapy likely to confer clinical benefit; or a participant who is not a candidate for such available therapy and for whom, in the opinion of the investigator, experimental therapy with acasunlimab or acasunlimab in combination with pembrolizumab may be beneficial.
* Asian race and Japanese ethnicity.
* Have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Have Eastern Cooperative Oncology Group (ECOG) 0-1.
* Have an acceptable hematological status.
* Have acceptable liver function.
* Have an acceptable coagulation status.
* Have acceptable renal function.
* Should provide a tumor tissue sample (formalin-fixed paraffin-embedded [FFPE] blocks/slides) from archival tissue or fresh biopsy collected before C1D1, preferably derived from advanced disease stage.

Key Exclusion Criteria:

* Have uncontrolled intercurrent illness, including but not limited to:

  * Ongoing or active infection requiring intravenous treatment with anti-infective therapy, or any ongoing systemic inflammatory condition requiring further diagnostic work-up or management during screening.
  * Symptomatic congestive heart failure (Grade III or IV as classified by the New York Heart Association), unstable angina pectoris or cardiac arrhythmia.
  * Uncontrolled hypertension defined as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg, despite optimal medical management.
  * Ongoing or recent evidence of autoimmune disease.
  * History of irAEs that led to prior checkpoint treatment discontinuation.
  * Prior history of myositis, Guillain-Barré syndrome, or myasthenia gravis of any grade.
  * History of chronic liver disease or evidence of hepatic cirrhosis.
  * Evidence of interstitial lung disease.
  * History of non-infectious pneumonitis that has required steroids or currently has pneumonitis.
  * History of organ allograft (except for corneal transplant) or autologous or allogeneic bone marrow transplant, or stem cell rescue within 3 months prior to the first dose of trial treatment.
  * Serious, non-healing wound, skin ulcer (of any grade), or bone fracture.
* Any history of intracerebral arteriovenous malformation, cerebral aneurysm, new (younger than 6 months) or progressive brain metastases or stroke.
* Prior therapy:

  * Radiotherapy: Radiotherapy within 14 days prior to the first dose of trial treatment. Palliative radiotherapy will be allowed.
  * Treatment with an anti-cancer agent (within 28 days or after at least 5 half-lives of the drug, whichever is shorter), prior to trial treatment administration.
* Toxicities from previous anti-cancer therapies that have not adequately resolved.

Note: Other protocol specified inclusion/exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose limiting Toxicities (DLTs) | During first cycle (Cycle length=21 days) in each cohort
  Determine the DLT profile of acasunlimab administered as monotherapy or in combination with pembrolizumab. The DLTs will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria version 5.0.
Number of Participants with Adverse Events (AEs) | From first dose date up to end of the safety follow up period, 90 days after last dose
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Area under the concentration time curve (AUC) of Acasunlimab | Predose and postdose at multiple timepoints of each cycle (Cycle length=21 days)
Maximum (Peak) Plasma Concentration (Cmax) of Acasunlimab | Predose and postdose at multiple timepoints of each cycle (Cycle length=21 days)
Time to Reach Cmax (Tmax) of Acasunlimab | Predose and postdose at multiple timepoints of each cycle (Cycle length=21 days)
Plasma Trough (Pre-dose) Concentrations (Cthrough) of Acasunlimab | Predose and postdose at multiple timepoints of each cycle (Cycle length=21 days)
Elimination half-life (t 1/2) of Acasunlimab | Predose and postdose at multiple timepoints of each cycle (Cycle length=21 days)

SECONDARY OUTCOMES:
Number of Participants with Anti-Drug Antibody (ADA) to Acasunlimab | Up to 2 years
  Serum samples will be screened for ADAs to acasunlimab and the titer of confirmed positive samples will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (2):
- Japan (2):
  - National Cancer Center East, Chiba
  - National Cancer Center Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No